CLINICAL TRIAL: NCT01345084
Title: A Phase III Study Evaluating the Standard Radiation Therapy and Chemotherapy Regimen, With or Without Nimotuzumab, in Unresectable, Locally Advanced Epidermoid Carcinoma of the Head and Neck
Brief Title: Study Comparing Radiation Therapy and Chemotherapy With or Without Nimotuzumab
Acronym: NICAP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: change company strategy
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF 118
Record Dates: First submitted 2011-04-28; First posted 2011-04-29 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2013-08

CONDITIONS: Carcinoma; Head and Neck Cancer
MeSH Terms: conditions — Carcinoma; Head and Neck Neoplasms | interventions — Radiotherapy; nimotuzumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiation therapy, cisplatin and nimotuzumab (Experimental): Nimotuzumab - (Diluted into 250 mL of sodium chloride sterile solution 0.9% in intravenous infusion for 30 minutes. Pre-drugs are optional, at the investigator's discretion)- 200 mg, IV, weekly doses during the radiation therapy until completing 6 months.
  Radiation therapy- 66 -70 Gy, external,fractions of 2 Gy per day, 5 days a week
  Cisplatin - 75 mg/m2, IV, Doses every 3 weeks (a total of three doses)
  Interventions: Drug: Nimotuzumab
- Radiation therapy and cisplatin (Active Comparator): Radiation therapy: 66- 70 Gy, fractions of 2 Gy per day, 5 days a week
  Cisplatin:75 mg/m2, IV, doses every 3 weeks (a total of three doses)
  Interventions: Radiation: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiation Therapy — 66- 70 Gy External, Fractions of 2.0 Gy per day, 5 days a week
  Arms: Radiation therapy and cisplatin
Drug: Nimotuzumab — 200 mg, IV, weekly doses during the radiation therapy until completing 6 months (Diluted into 250 mL of sodium chloride sterile solution 0.9% in intravenous infusion for 30 minutes).
  Arms: Radiation therapy, cisplatin and nimotuzumab
Drug: Cisplatin — 75 mg/m2, IV, doses every 3 weeks (a total of three doses)
  Arms: Radiation therapy and cisplatin

SUMMARY:
Primary: to compare the overall survival defined as the time elapsed between the randomization date and death due to any cause, in both treatment groups.

Secondary: to compare the progression-free survival, incidence of locoregional failure, site of the first recurrence/progression, objective response rate assessment, quality of life assessment and incidence of adverse events.

DETAILED DESCRIPTION:
This is a phase III, superiority, national, open-label, randomized, and two-arm study.

Patients' enrollment will be performed only after approval by competent regulatory authorities and it will last up to 12 months.

All patients taking part in the study must sign an informed consent. The patients will have stage III or IV, unresectable head and neck SCC, performance status 0 or 1.

Randomization and treatment assignment will be performed by a company specifically contracted for such purpose and will be per research site and disease stage, 1:1

ELIGIBILITY:
Inclusion Criteria

* Aged 18 to 75 years old;
* Histological or cytological confirmation of SCC in oral cavity, oropharynx, hypopharynx, or larynx;
* Stages III or IV disease
* Unresectability according to responsible surgeon or medical staff's opinion;
* Performance status 0 or 1
* Present indication for radiation therapy and chemotherapy treatment with cisplatin;
* Adequate hepatic, renal and medullar functions, indicated by:
* Life expectancy above 6 months.

Exclusion Criteria

* Presence of nasopharyngeal, paranasal sinuses, or salivary glands carcinoma;
* Presence of known distant metastasis;
* Presence of any other active neoplasm or history of any tumor diagnosed in the last 5 years
* Patients with inability to eat normally, in whom a gastric or enteral tubing was not possible at least 2 weeks before their enrollment in the study;
* Previous treatment with chemotherapy, radiation therapy, or EGFR inhibitors of any pharmacological class;
* Presence of serious comorbidity that, in the investigator's opinion, will put the patient at risk or will jeopardize protocol compliance;
* Active known seropositivity for HIV, hepatitis B or C
* Presence of a significant neurological or psychiatric disease, as per the investigator's judgment;
* Hypersensitivity or allergy to any of the study treatments;
* Presence of uncontrolled hypercalcemia;
* Pregnancy or breastfeeding;
* Female patients of childbearing potential who wish to become pregnant or are unwilling, as well as their partners, to use an appropriate contraceptive method throughout the study period;
* Participation in any clinical trial in the last 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6 months
  Local control of disease will be measured by magnetic resonance imaging (MRI) and physical examination 6 weeks after treatment end.

SECONDARY OUTCOMES:
Complete clinical response rate | 2 years
  Progression-free survival; Incidence of locoregional failure; Site of the first recurrence or progression; Objective response rate assessment; EORTC quality of life questionnaires assessment; Incidence of several adverse events;

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Girotto, Principal Investigator — Hospital de Base São José do Rio Preto
Locations (8):
- Brazil (8):
  - Hospital Erasto Gaetner, Curitiba, Paraná
  - Hospital Federal de Bonsucesso, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Centro Oncológico de Mogi das Cruzes, Mogi das Cruzes, São Paulo
  - Hospital de Base São José do Rio Preto, São José do Rio Preto, São Paulo
  - Instituto do Câncer de São Paulo, São Paulo, São Paulo